CLINICAL TRIAL: NCT03913936
Title: Young, Empowered & Strong (YES): The Young Women's Breast Cancer Study 2- Focus on Intervention Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-641
Record Dates: First submitted 2019-02-19; First posted 2019-04-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NEWLY DIAGNOSED (Experimental): Participants will track their symptoms with weekly and monthly standard surveys to monitor for symptoms.
  The YES portal is designed to collect and assess participants' toxicities and symptoms, as well as informational needs in between visits with their clinician
  Interventions: Other: YES portal
- SURVIVOR (Experimental): * Participants will track their symptoms with weekly and monthly standard surveys to monitor for symptoms.
  * The YES portal is designed to collect and assess participants' toxicities and symptoms, as well as informational needs in between visits with their clinician
  Interventions: Other: YES portal
- LIVING WITH ADVANCED DISEASE (Experimental): * Participants will track their symptoms with weekly and monthly standard surveys to monitor for symptoms.
  * The YES portal is designed to collect and assess participants' toxicities and symptoms, as well as informational needs in between visits with their clinician
  Interventions: Other: YES portal

INTERVENTIONS:
Other: YES portal — The YES portal is designed to collect and assess participants' toxicities and symptoms, as well as informational needs in between visits with their clinician

SUMMARY:
This research study is piloting a new internet-based research tool (YES portal). The main purpose of this pilot study is to test the web-based interface.

DETAILED DESCRIPTION:
This study is being done to pilot a web-based research intervention tool. The investigators hope that by piloting it with the participants they can improve the tool and the other processes. The main purpose of this pilot study is to test the web-based interface, the participant's engagement with the platform, and the recruitment procedures. This initial pilot study will inform the design of a larger study intended to monitor common symptoms and behavior, and to provide supportive care information and research opportunities in an iterative manner for young women who have been diagnosed with breast cancer using the YES portal, built for smartphones, tablets, and computers.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the ages of 18-44 years
* A history of breast cancer; we will pilot in 3 separate cohorts consisting of 10 patients each: newly diagnosed patients receiving care at DFCI, prevalent survivors who have completed early active therapy (surgery, chemotherapy and/or radiotherapy) and are being followed at DFCI, and women living with advanced breast cancer receiving care at DFCI
* Be fluent in and able to read English
* Have internet access on a regular basis at the time of consent that can support the web-based platform

Exclusion Criteria:

N/A

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Frequency of logging into the portal. | 2 years
  To measure the number of times participants engage with the portal using log in data collected from back-end of portal.
Time spent in the portal. | 2 years
  To summarize the number of hours/minutes the participant spent using portal through data collected from back-end of portal.
Time spent responding the survey. | 2 years
  To summarize the number of hours/minutes the survey takes to complete through data collected from back-end of portal.
Frequency of information downloads. | 2 years
  To measure the number of times participants download the resource sources provided through data collected from back-end of portal.
Participant-reported utility of the portal. | 2 years
  Investigator developed questions will be used to assess the utility of the portal including the perceived usefulness of portal in addressing symptoms and needs and ease of use.
Participant-reported recommendations for improving the portal. | 2 years
  Investigator developed questions asking participants for feedback pertaining to ways to improve the portal and processes.

CONTACTS AND LOCATIONS:
Overall Officials: Ann H. Partridge, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation
URL: https://www.dana-farber.org/research/innovations